CLINICAL TRIAL: NCT02614209
Title: A Blood Collection From Patients Presenting in the Emergency Department and Prescribed a Brain Natriuretic Peptide (BNP) Laboratory Test
Brief Title: Blood Collection of Patient Presenting in the ED and Prescribed a BNP
Acronym: BNP
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-120
Record Dates: First submitted 2015-11-06; First posted 2015-11-25 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: ED; BNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: In Vitro diagnostic tests — Prospective blood collection
  Other Names: Propective collection for use in InVitro diagnostic studies

SUMMARY:
Plasma specimen collected from patients presenting in the Emergency Department (ED) with or without Heart Failure (HF) and prescribed a BNP.

DETAILED DESCRIPTION:
Plasma samples are collected from a minimum of 400 subjects. Specimens are used to confirm the currently accepted BNP cut off as and aid in the diagnosis and assessment of HF.

Stored specimens for future use in BNP assay development.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >21 years of age
* Able to understand and willing to provide informed consent
* Present in to ED
* BNP test requested

Exclusion Criteria:

* Males and females< 21 years
* Unable to provide informed consent
* Not presenting to ED
* hemolyzed sample

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to ED and prescribed a BNP with or without HF
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Measure BNP | 6 months
  400 subjects

CONTACTS AND LOCATIONS:
Overall Officials: Diana Dickson, RAC, Study Director — Fujirebio Diagnostics, Inc.
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan